CLINICAL TRIAL: NCT06353152
Title: An Early Exploratory Clinical Trial of Claudin18.2-Targeted Chimeric Antigen Receptor T Cell Therapy for Gastric/Gastroesophageal Junction Adenocarcinoma.
Brief Title: Claudin 18.2-Targeted Chimeric Antigen Receptor T-cells for Gastric/Gastroesophageal Junction Adenocarcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: Gracell Biopharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Shen Lin, Principal Investigator, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC506-507
Record Dates: First submitted 2023-11-15; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Claudin18.2-Targeted Chimeric Antigen Receptor T Cell Injection (Experimental): The subjects enrolled will be sequentially assigned to the corresponding dose level.
  Interventions: Drug: Claudin18.2-Targeted Chimeric Antigen Receptor T Cell Injection

INTERVENTIONS:
Drug: Claudin18.2-Targeted Chimeric Antigen Receptor T Cell Injection — single-/multiple-dose infusion

SUMMARY:
A single-arm, open-label early-stage exploratory clinical study to evaluate the safety, tolerability and efficacy of Claudin 18.2-Targeted Chimeric Antigen Receptor T-cells in subjects with gastric/gastroesophageal junction adenocarcinoma.

DETAILED DESCRIPTION:
This study is an open-label, single-/multiple-dose infusion, adaptive dose-escalation designed early exploratory clinical trial aiming to evaluate the safety, tolerability, and efficacy of Claudin18.2-Targeted Chimeric Antigen Receptor T Cell Injection in subjects with CLDN18.2 positive and pathologically confirmed locally advanced or metastatic gastric/gastroesophageal junction adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-70 years old (including the threshold);
2. Subject has pathologically confirmed locally advanced or metastatic gastric/gastroesophageal junction adenocarcinoma：Having received at least one standard treatment, with the disease in stable or progressive state, and the subject refusing further treatment or intolerant to existing therapies; Failing second-line treatment;
3. Subject's freshly biopsied tumor tissue (if the patient has not received targeted Claudin18.2 therapy, archived tumor tissue within one year is acceptable) has immunohistochemistry confirmed positive expression of Claudin18.2;
4. Subject has predicted life expectancy ≥ 90 days;
5. Subject has Eastern Cooperative Oncology Group (ECOG) performance status 0-1;
6. Subject is willing to undergo tumor biopsy;
7. Subject has at least one measurable tumor lesion on imaging (per RECIST 1.1 criteria);
8. Female subjects of childbearing age must not be lactating, and sensitive serum pregnancy test during the screening period must be negative for fertile women. All subjects must use medically accepted contraceptive measures (such as intrauterine devices, contraceptives) throughout the treatment period and 1 year after cell infusion. Male subjects must also avoid sperm donation;
9. Subject has adequate organ function reserves: Absolute neutrophil count (ANC) ≥ 1.5×109/L; Absolute lymphocyte count (ALC) ≥ 0.6×109/L; Platelet count ≥ 75×109/L; Hemoglobin ≥ 9.0 g/dL; Total bilirubin ≤ 2 × upper limit of normal (ULN) ; ALT and AST ≤ 2.5 × ULN (or ≤ 5 × ULN if bone or liver metastases are present); Creatinine clearance (Cockcroft-Gault method) ≥ 60 mL/min; Stable coagulation function: Prothrombin time (PT) ≤ 1.5 × ULN; Activated partial thromboplastin time (APTT) ≤ 1.5 × ULN; Echocardiography shows left ventricular ejection fraction (LVEF) ≥ 55% without moderate or severe pericardial effusion; Baseline oxygen saturation in room air ≥ 92%;
10. Subject is able to establish intravenous access, and peripheral blood mononuclear cells can be collected according to the investigator's judgment;
11. Subject is willing to sign the informed consent form;
12. Subject can communicate well with the investigator, is willing and able to comply with the study plan and will complete the study as per the study requirements.

Exclusion Criteria:

1. Subject has a positive test for Hepatitis B surface antigen (HBsAg) or Hepatitis C virus antibody (HCV-Ab) or Treponema pallidum antibody (TP-Ab) or Human Immunodeficiency Virus antibody (HIV-Ab). Subjects who are positive for both hepatitis B core antibody (HBcAb) and HBV deoxyribonucleic acid (DNA) will be excluded.
2. Subject has other malignant tumors, except for: cured non-melanoma skin cancer, in situ cervical carcinoma, localized prostate cancer, superficial bladder cancer, ductal carcinoma in situ, and other malignant tumors with disease-free survival exceeding 5 years.
3. Subject has symptomatic intracranial metastases.
4. Subject has central or extensive lung or liver metastases.
5. Subject with a maximum target lesion > 4.0 cm (per RECIST 1.1 criteria).
6. The subjects' tumor tissue is positive for HER2 expression.
7. Subject has a history of prior anti-tumor treatment or participation in clinical trials: subject has received treatment with CAR-T therapy, or other gene-edited cell therapies; subject has participated in other clinical trials within 28 days before screening; Subject has received local radiotherapy or small molecule chemotherapy within 7 days before leukapheresis, or within at least five half-lives (whichever is longer).; subject has received daily systemic corticosteroid ≥ 15 mg within 7 days before leukapheresis, except inhaled corticosteroids.
8. Subject has received vaccination within 28 days before screening.
9. Subject has conditions requiring the use of systemic corticosteroids or other immunosuppressive drugs during the study period, as determined by the investigator.
10. Subject has acute toxic reactions from previous treatments not recovered to Grade 1 or lower (excluding hematological toxicity, alopecia, and events considered tolerable by the investigator).
11. Subject has life-threatening hypersensitivity reactions or other intolerances to cyclophosphamide, fludarabine, or albumin-bound paclitaxel, or severe hypersensitivity to human serum albumin, DMSO, or other substances.
12. Subject underwent general anesthesia within 28 days before screening, or has not recovered and clinically stabilized after previous surgical treatment, or is expected to undergo general anesthesia during the study.
13. Subject has any unstable cardiovascular diseases within 180 days before screening, including but not limited to unstable angina, myocardial infarction, heart failure (New York Heart Association [NYHA] class ≥ III), severe arrhythmias requiring medication, or underwent cardiovascular intervention, coronary artery stenting, or coronary artery bypass grafting within 180 days before screening.
14. Subject has a disease or history of central nervous system disorders, such as epilepsy, cerebral ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune diseases involving the CNS.
15. Subject has uncontrolled or requiring intravenous treatment for fungal, bacterial, viral, or other infections at the time of screening.
16. Subject has uncontrolled or active ulcers or gastrointestinal bleeding at the time of screening.
17. Subject has active autoimmune diseases (including but not limited to systemic lupus erythematosus, Sjögren's syndrome, rheumatoid arthritis, psoriasis, multiple sclerosis, inflammatory bowel disease, Hashimoto's thyroiditis, etc., with the exception of hypothyroidism that can be controlled only by hormone replacement therapy).
18. Subject has a bleeding and thrombotic tendency, including: subject who had significant clinically significant bleeding symptoms or definite bleeding tendencies within 90 days before screening, subject who has genetic or acquired bleeding and thrombotic tendencies (e.g., hemophilia, coagulation disorders, splenic hyperfunction), subject who is undergoing thrombolysis or anticoagulant therapy and subject who had events of arterial/venous thrombosis within 180 days before screening, such as cerebrovascular disease (including cerebral hemorrhage, cerebral infarction), deep venous thrombosis, and pulmonary embolism.
19. Subject has a history of substance abuse with psychiatric drugs and unable to abstain, or with a history of psychiatric disorders.
20. Subject has other situations in which the investigator deems unsuitable for participation in this clinical study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2025-11-16 (Estimated); Study Completion 2025-11-16 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Dose limiting toxicity. | Within 28 days after the first infusion
  Occurrence of DLTs (Dose limiting toxicity).
Incidence of treatment-emergent AEs, AESIs, and SAEs. | 48 weeks
  Incidence of treatment-emergent AEs, AESIs, and SAEs.

SECONDARY OUTCOMES:
Disease control rate (DCR) | 12 months
  The proportion of participants who have a confirmed CR, confirmed PR, or who have SD per RECIST v1.1 as assessed by the investigator at local site and derived from the raw tumor data for at least 11 weeks after infusion date.
Objective response rate (ORR) | 12 months
  The proportion of participants who have a confirmed CR or confirmed PR as determined by the investigator at local site per RECIST v1.1.
Duration of disease control (DDC) | 12 months
  The period from the first evaluation of CR, PR or SD to the first evaluation of PD or any cause of death.
Duration of response (DOR) | 12 months
  The period from the first evaluation of CR or PR to the first evaluation of PD or death of any cause.
Progression-free survival (PFS) | 12 months
  The period from the first cells infusion to the first recorded tumor progression or death of any cause.
Overall survival (OS) | 12 months
  The period from the first cells infusion to death of any cause.
Proliferation and persistence of Claudin18.2-Targeted Chimeric Antigen Receptor T Cell | 12 months
  Proliferation and persistence of Claudin18.2-Targeted Chimeric Antigen Receptor T Cell Injection in peripheral blood after infusion detected by Quantitative Real-time PCR (qPCR) and Flow Cytometry (FCM).
Incidence of anti-CAR-T cell antibody in peripheral blood after infusion. | 12 months
  Incidence of anti-CAR-T cell antibody in peripheral blood after infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, PHD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No